CLINICAL TRIAL: NCT06317714
Title: Non-interventional and Longitudinal Study to Evaluate a List of Anticancer Drugs Under Real Conditions of Use and Measure the Quality of Life of Patients Treated at Rafaël Institute
Brief Title: Long-term Follow-up and Quality of Life of Patients Treated With Anticancer Drugs
Acronym: THERAPINNOV
Status: Recruiting | Type: Observational
Sponsor: Institut Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: IR-2023/0002; 2023-A02233-42 (Other: ANSM)
Record Dates: First submitted 2024-03-08; First posted 2024-03-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Oncology; Quality of Life; Symptoms and Signs
MeSH Terms: conditions — Neoplasms; Signs and Symptoms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — o Quality of life questionnaires EORTC QLQC-30 and EQ-5D-5L
  ° questionnaires NCI- PRO-CTCAE

SUMMARY:
Currently, aspects related to the effects of anticancer treatments and the quality of life of patients and their needs are still poorly documented at the Rafael Institute. Thus this study will meet a dual objective: (1) the establishment of a registry to collect data on the safety and effectiveness of innovative and expensive anticancer drugs when administered in real life and (2) a measurement quantitative quality of life of patients treated with these drugs.

DETAILED DESCRIPTION:
In France, the promotion of more patient-centered medicine is among the priorities identified by the High Authority for Health in its 2024 strategic project. The patient-centered approach is based on a partnership relationship with the patient, their loved ones, and the healthcare professional or a multi-professional team to built together the best option of care.

In this approach, the Rafael Institute was created with the objective of caring for people and not simply pathologies. Initiated around the problem of cancer and the harmful effects of its treatments, the Rafaël Institute offers personalisation of care and continuity of care over time by providing monitoring and support to the patient by a multi-professional and multidisciplinary team. Thus, maintaining quality of life constitutes one of the objectives of the therapeutic management of patients with cancer.

Although modern oncological treatments have today enabled real advances on the biomedical level, they often have side effects that must be taken into account for the overall assessment and management of patients. Although most anticancer therapies have a negative impact on the patient's quality of life, this does not always reflect the occurrence of toxicity.

Since the 1990s, quality of life has been strongly associated with survival. Patients with high overall quality of life live significantly longer than patients with low overall quality of life.

The relationship between symptoms, their intensity and quality of life is essential to study to understand the perceived impact of treatments and optimize their use in daily practice.

The effects of treatment and quality of life can be assessed precisely and reliably using standardized and validated self-questionnaires. Completed by patients, they make it possible to measure the qualitative aspects directly linked to their health and to take into account their subjective perception of their state of health.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years (adult)
* Patients treated with an anticancer drug included in the list of innovative/expensive therapies (protocol appendix)
* Patients benefiting from non-pharmacological treatment at the Rafael Institute
* Who understands the French language

Exclusion Criteria:

* < 18 years old
* Patient deprived of liberty, under guardianship or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Rafael Institute for whom treatment with an anticancer drug (innovative/expensive molecule from the list annexed to the protocol) has been indicated.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | Until death, assessed up to 36 months
  OS is defined as the time from the starting date of study drug to the date of death due to any cause.
progression free survival | Until progression or death, assessed up to 36 months
  PFS is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first.
incidence of adverse events | up to 36 months
  graded according to NCI CTCAE v5.0
incidence of serious adverse events | up to 36 months
  graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Change from Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Questionnaire Core 30 (QLQ-C30) Score | every 6 months and up to 36 months
  The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Individual responses for each of 28 items are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome, and responses for each of 2 items (overall health and overall quality of life) are given on a 7-point scale (1=Very poor to 7=Excellent), with a higher score indicating a better outcome.
change from baseline in quality of life measured with the EQ5D5L questionnaire | every 6 months and up to 36 months
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. The levels of severity for each dimension ranges from no problems (1) to extreme problems/unable to perform. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Rafaël, Levallois-Perret, Institut Rafael, France

IPD SHARING:
Plan to Share IPD: No